CLINICAL TRIAL: NCT05235789
Title: Evaluation of Individual Intervention With Rational Emotional Behavioral Therapy Performed by Primary Care Clinical Social Workers in People With a New Episode of Depression: a Randomized Clinical Trial
Brief Title: Cognitive Behavioral Therapy (REBT) Evaluation for Depression at Primary Care.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Català de la Salut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21/152-P
Record Dates: First submitted 2021-12-13; First posted 2022-02-11 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Depression
Keywords: Effectiveness; cost effectiveness; rational behavioral emotional therapy; depression; clinical trial
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with control group, in people diagnosed with major depression attached to the PC.
  This study is carried out in 9 primary care centers in Catalonia.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The social workers in each center of primary care held eight 30 minutes sessions fortnightly of Rational-Emotive-Behavioral Therapy. First session is informative about the type of treatment to be performed. The next sessions work events, thoughts and feelings with the goal of changing the dysfunctional thoughts by other more rational ones, measured by scales.
  Interventions: Other: Rational-Emotive-Behavioral Therapy
- Control group (Active Comparator): The control group (GC) in each center of primary care will take the usual medical care for depression, according with up-dated national and international guidelines.
  Interventions: Other: Control Group usual care

INTERVENTIONS:
Other: Rational-Emotive-Behavioral Therapy — The structure of the REBT sessions includes the following points:
  1. Determine specific goals that explain what the participant want to achieve through the content of the session.
  2. Explain the level of skills to be achieved in each session.
  3. Development of the session, reminder of the previous session, review of homework (from the second session to the 8th). Irrational beliefs and disruptive thoughts will be worked on together with the participant in order to achieve an improvement in their emotional state. Key messages with healthier alternatives that make your daily life easier.
  4. Establishing homework. Using the REBT Toolbox with Key Messages.
  5. Individual psychosocial work will be recorded in the computerized medical history.
  Other Names: Cognitive-Emotive-Behavioral Therapy; REBT; CBT; REBT-CBT
  Arms: Intervention group
Other: Control Group usual care — In the control group, for each center , the depression is treated as usual with the conventional treatment, according to national and international guidelines.
  Other Names: conventional treatment; usual care
  Arms: Control group

SUMMARY:
Background: Rational Emotional Behavioral Therapy (REBT) applied by the Primary Health Care (PC) Social Worker reduces psychotropic drug use and overcrowding at medical appointments.

Hypothesis: The REBT in people diagnosed with mild-moderate depression in the social work consultation of PC, improves the clinical control of this disorder, with lower consumption of health resources, better quality of life and user satisfaction, with respect to the usual clinical practice, in addition to being cost-effective.

Goals: To compare the effectiveness, cost-effectiveness and cost-utility of REBT as an intervention tool with respect to the usual clinical practice in adults with a diagnosis of mild-moderate major depression in PC.

Methodology: Randomized clinical trial with control group, in people diagnosed with major depression attached to the PC. This study is carried out in 9 primary care centers in Catalonia.

Determinations: Participants are measured at the beginning of the study, end of the intervention and at 1 year of the beginning: Control of symptoms using PHQ-9; Health-related quality of life using the EQ-5D-5L scale; Self-perceived well-being, using the Ryff Psychological Well-Being Scale; Pharmacological prescription and withdrawal of anxiolytics, hypnotics and antidepressants; Frequency of PC consultations; Assignable costs through TIC-P; Functional social support perceived prior to the intervention using the Duke questionnaire; and user satisfaction with the treatment at the end of the intervention using CRES-4.

The exposure variable is the assignment to the REBT psychosocial intervention group or the usual clinical practice control group.

Statistical analysis: Description of the items of the measuring instruments used per month will calculate the cost by variation of quality-adjusted life year (QALY) and the increase of associated cost-effectiveness ratio contrasting the hypothesis that this is different to 22000 € by means of t-test.

Expected results: REBT in people diagnosed with mild-moderate depression in the social work consultation of PC, will improve in the clinical control of this disorder, a lower consumption of health resources, improvement in the Quality of Life and in the user satisfaction. Therefore, REBT is effective, and cost-effective in managing people diagnosed with mild-moderate major depression.

Applicability and Relevance: REBT will help people to acquire tools to deal with difficulties in daily life and provide economic savings in health care costs.

ELIGIBILITY:
Inclusion Criteria:

Patients treated at the primary care medical consultation , who signed the Informed Consent, with:

* first diagnosis of mild (F32.0)
* moderate major depression (F32.1, F32.9 (unspecified depression).

Exclusion Criteria:

* Participants diagnosed with severe depression F32.2, psychotic major depression F32.3, moderate recurrent depression F33.1, severe recurrent depression F33.2 or Beck test> 30 points at baseline visit
* Any other type of psychiatric pathology (F60.9 personality disorder, F20.9 schizophrenia, F42.9 obsessive compulsive disorder, F20.0 paranoid schizophrenia, F31.9 bipolar disorder, F43.10 post-traumatic stress disorder, obsessive compulsive disorder F42.9.
* Impaired cognitive ability according to PFEIFFER SPMSQ Scale (Short Portable Mental State Questionnaire) (<3 points)
* Dementia - presenile dementia - senile dementia (F03.90). All three share code, dementia Sclerotic artery - vascular dementia - multiinfarct dementia (F01.50). All three share code. Alzheimer's disease (G30) and Lewy body dementia (G31.89)
* Person included in home care (Z74.9)
* The unwillingness to treat.
* Participation in psychoeducational groups of the Catalan Institute of Health ("Institut Català de la Salut" -ICS-), or other individual or group psychological therapies.
* Any pathology or circumstance that makes it impossible for the user to participate in the study and / or the follow-up required by the same:
* Terminal illnesses, (life expectancy of less than one year according to ECAP); Advanced Chronic Diseases (MACA in the section on chronicity in the ECAP)
* Illiteracy and / or language barrier
* Deaths and transfers from the generation of the recruitment list from the beginning of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | It will be measured as baseline.
  The PHQ-9 questionnaire consists of 9 items that assess the presence of depressive symptoms (corresponding to Diagnostic and Statistical Manual of Mental Disorders -DSM-IV-) in the last 2 weeks, according to frequency: 0 = "never", 1 = "some days", 2 = "more than half the days "and 3 =" almost every day "; allows a classification in "Major Depressive Syndrome", "Other Depressive Syndromes", "Positive Depressive Symptoms" or "Negative Depressive Symptoms". However, in the present study we will use the total score (unweighted summation of item scores) as a measure of depressive symptoms.
Patient Health Questionnaire (PHQ-9) | It will be measured at 4 months from baseline.
  The PHQ-9 questionnaire consists of 9 items that assess the presence of depressive symptoms (corresponding to Diagnostic and Statistical Manual of Mental Disorders -DSM-IV-) in the last 2 weeks, according to frequency: 0 = "never", 1 = "some days", 2 = "more than half the days "and 3 =" almost every day "; allows a classification in "Major Depressive Syndrome", "Other Depressive Syndromes", "Positive Depressive Symptoms" or "Negative Depressive Symptoms". However, in the present study we will use the total score (unweighted summation of item scores) as a measure of depressive symptoms.
Patient Health Questionnaire (PHQ-9) | It will be measured at 1 year from baseline.
  The PHQ-9 questionnaire consists of 9 items that assess the presence of depressive symptoms (corresponding to Diagnostic and Statistical Manual of Mental Disorders -DSM-IV-) in the last 2 weeks, according to frequency: 0 = "never", 1 = "some days", 2 = "more than half the days "and 3 =" almost every day "; allows a classification in "Major Depressive Syndrome", "Other Depressive Syndromes", "Positive Depressive Symptoms" or "Negative Depressive Symptoms". However, in the present study we will use the total score (unweighted summation of item scores) as a measure of depressive symptoms.
5-Dimensional, 5-Level EuroQol Questionnaire (EQ-5D-5L) | It will be measured as baseline.
  The EuroQol 5D5L questionnaire contains an Analog Visual Scale, and 5 items / dimensions (mobility, personal care, daily activities, pain / discomfort and anxiety / depression), rated at 5 levels ("No problems", "mild problems", "moderate problems", "severe problems" and "extreme problems or incapable of") . The final profit index will be calculated using the standardized hybrid method (compound time equivalence / discrete choice experiments) of Spanish social preferences.
5-Dimensional, 5-Level EuroQol Questionnaire (EQ-5D-5L) | It will be measured at 4 months from baseline.
  The EuroQol 5D5L questionnaire contains an Analog Visual Scale, and 5 items / dimensions (mobility, personal care, daily activities, pain / discomfort and anxiety / depression), rated at 5 levels ("No problems", "mild problems", "moderate problems", "severe problems" and "extreme problems or incapable of") . The final profit index will be calculated using the standardized hybrid method (compound time equivalence / discrete choice experiments) of Spanish social preferences.
5-Dimensional, 5-Level EuroQol Questionnaire (EQ-5D-5L) | It will be measured at 1 year from baseline.
  The EuroQol 5D5L questionnaire contains an Analog Visual Scale, and 5 items / dimensions (mobility, personal care, daily activities, pain / discomfort and anxiety / depression), rated at 5 levels ("No problems", "mild problems", "moderate problems", "severe problems" and "extreme problems or incapable of") . The final profit index will be calculated using the standardized hybrid method (compound time equivalence / discrete choice experiments) of Spanish social preferences.
Scale of Psychological Well-Being (Ryff, 1989). | It will be measured as baseline.
  Reduced self-perceived well-being questionnaire of 29 items, subdivided into 6 dimensions with statements about Self-Acceptance, Positive Relationships, Autonomy, Mastery of the Environment, Personal Growth and Purpose in Life. It uses a 6-point likert scale where 1 strongly agrees and 6 strongly disagrees. The final results will be by dimensions.
Scale of Psychological Well-Being (Ryff, 1989). | It will be measured at 4 months from baseline.
  Reduced self-perceived well-being questionnaire of 29 items, subdivided into 6 dimensions with statements about Self-Acceptance, Positive Relationships, Autonomy, Mastery of the Environment, Personal Growth and Purpose in Life. It uses a 6-point likert scale where 1 strongly agrees and 6 strongly disagrees. The final results will be by dimensions.
Scale of Psychological Well-Being (Ryff, 1989). | It will be measured at 1 year from baseline.
  Reduced self-perceived well-being questionnaire of 29 items, subdivided into 6 dimensions with statements about Self-Acceptance, Positive Relationships, Autonomy, Mastery of the Environment, Personal Growth and Purpose in Life. It uses a 6-point likert scale where 1 strongly agrees and 6 strongly disagrees. The final results will be by dimensions.
Treatment Inventory Cost in Psychiatric patients (TIC-P) | It will be measured as baseline.
  The TIC-P questionnaire includes 8 general questions, costs in two dimensions: use of health resources (direct costs, 35 questions) and loss of productivity (indirect costs, Institute for Medical Technology Assessment (iMTA) Productivity Cost Questionnaire -iPCQ-, 12 questions).
Treatment Inventory Cost in Psychiatric patients (TIC-P) | It will be measured at 4 months from baseline.
  The TIC-P questionnaire includes 8 general questions, costs in two dimensions: use of health resources (direct costs, 35 questions) and loss of productivity (indirect costs, Institute for Medical Technology Assessment (iMTA) Productivity Cost Questionnaire -iPCQ-, 12 questions).
Treatment Inventory Cost in Psychiatric patients (TIC-P) | It will be measured at 1 year from baseline.
  The TIC-P questionnaire includes 8 general questions, costs in two dimensions: use of health resources (direct costs, 35 questions) and loss of productivity (indirect costs, Institute for Medical Technology Assessment (iMTA) Productivity Cost Questionnaire -iPCQ-, 12 questions).
Attendance of primary care during the previous year. | It will be measured as baseline.
  Number of scheduled PC visits (both face-to-face and telephone) for physician / social worker / nurse, in the year prior to the start of the study, and at the end of follow-up.
Attendance of primary care during the previous year. | It will be measured at baseline.
  Number of scheduled PC visits (both face-to-face and telephone) for physician / social worker / nurse, in the year prior to the start of the study, and at the end of follow-up.
Attendance of primary care during the previous year. | It will be measured at 1 year from baseline.
  Number of scheduled PC visits (both face-to-face and telephone) for physician / social worker / nurse, in the year prior to the start of the study, and at the end of follow-up.
Duke Functional Social Support Questionnaire. | It will be measured at 4 months from baseline.
  The Duke Functional Social Support Questionnaire consists of 11 Likert-type items from 1 ("much less than I want") to 5 ("as much as I want"). It measures perceived social support and has two dimensions: "confidential social support" and "affective social support".
Satisfaction Scale with the treatment received (CRES-4). | It will be measured at 4 months from baseline.
  The CRES-4 scale measures 4 items likert: satisfaction with treatment (rated 0-5; "completely dissatisfied" and "completely satisfied, respectively), degree of resolution (0-5), previous emotional state (0-4), current emotional state (0-4). Three dimensions are derived from 0 (worst rating) to 100 (best rating): satisfaction, problem solving, and perception of emotional change.

CONTACTS AND LOCATIONS:
Overall Officials: Carme Rovira Aler, LCSW, Principal Investigator — Catalan Institute of Health
Locations (1):
- Catalan Health Institute. ABS Sant Andreu 9D, Barcelona, Spain